Table 3. The Distribution of Total Scale Score on the perpective of HLSBS II and its Sub-Dimensions Before and After Training in Group and Between Groups (n=128)

| Sub-Dimention of Scale | Intervention Group (n=63) | | Control Group (n=65) | | |
|---|---|---|---|---|---|
| | X±SS | Median-Min.Max. | X±SS | Median-Min.Max. | Analysis** (Intergroup) |
| Negative Impact. Somatic complaints BT. | 2.66 ± 0.83 | 2.38 (1.46-4.69) | 2.72± 0.91 | 2.69 (1-4.69) | t=0.392 p=0.696 |
| Negative Impact. Somatic complaints AT. | 2.35 ± 0.67 | 2.31 (1.23-4) | 2.80± 0.86 | 2.85 (1-4.54) | t=3.278 <b>p=0.001</b> |
| | t=4.8 | 06 <b>p&lt;0.001</b> | t=-0.875 p=0.385 | | |
| Pain Symptoms BT. | 3.11± 0.96 | 3.33 (1.17-4.83) | 2.99± 1.09 | 3.17 (1-5) | t=-0.643 p=0.522 |
| Pain Symptoms AT. | 2.57±0.75 | 2.50 (1.33-4.83) | 3.04± 1.16 | 3.00 (1-5) | t=2.676 p= <b>0.009</b> |
| | t=6.9 | 90 <b>p&lt;0.001</b> | t=- | 0.451 p=0.654 | |
| Coping Methods BT. | 2.38± 1.13 | 2.33 (1-5) | 2.24 <b>±</b> 1.14 | 2.00 (1-5) | t=-0.699 p=0.486 |
| Coping Methods AT. | 2.35± 0.94 | 2.33 (1-5) | 2.23± 1.16 | 2.00 (1-5) | t=-0.636 p=0.526 |
| | t=0.2 | 95 p=0.769 | p=0.963 | | |
| MSS BT. | 2.74± 0.77 | 2.59 (1.5-4.5) | 2.73± 0.89 | 2.59 (1-4.77) | t=-0.101 p=0.919 |
| MSS AT. | 2.41± 0.63 | 2.27 (1.36-3.91) | 2.79± 0.88 | 2.77 (1.05-4.68) | t=2.761p= <b>0.007</b> |
| Analysis* (in-group) | t=5.8 | 98 <b>p&lt;0.001</b> | t=-0. | 728 p=0.470 | |

**Table 4.** The Distribution of Total Scale Score related to MSQ and its Sub-Dimensions Before and After Training in Group and Between Groups (n=128).

| Sub-Dimention of Scale | Intervention (n=63) | | Control (n=65) | | Analiz** |
|---|---|---|---|---|---|
| | N±SS | Median-Min.Mak. | X±SS | Median-Min.Mak. | (Intergroup) |
| Negative Impact. Somatic complaints BT. | 2.66 ± 0.83 | 2.38 (1.46-4.69) | 2.72± 0.91 | 2.69 (1-4.69) | t=0.392 p=0.696 |
| Negative Impact. Somatic complaints AT. | 2.35 ± 0.67 | 2.31 (1.23-4) | 2.80± 0.86 | 2.85 (1-4.54) | t=3.278 <b>p=0.001</b> |
| | t=4.806 <b>p&lt;0.001</b> | | t=-0.875 p=0.385 | | |
| Pain Symptoms BT. | 3.11± 0.96 | 3.33 (1.17-4.83) | 2.99± 1.09 | 3.17 (1-5) | t=-0.643 p=0.522 |
| Pain Symptoms AT. | 2.57±0.75 | 2.50 (1.33-4.83) | 3.04± 1.16 | 3.00 (1-5) | t=2.676 p= <b>0.009</b> |
| | t=6.990 <b>p&lt;0.001</b> | | t=-0.451 p=0.654 | | |

| Coping Methods BT. | 2.38± 1.13 | 2.33 (1-5) | 2.24± 1.14 | 2.00 (1-5) | t=-0.699 p=0.486 |
|---|---|---|---|---|---|
| Coping Methods AT. | 2.35± 0.94 | 2.33 (1-5) | 2.23± 1.16 | 2.00 (1-5) | t=-0.636 p=0.526 |
| | t=0.295 p=0.769 | | t=0.046 p=0.963 | | |
| MSS BT. | 2.74± 0.77 | 2.59 (1.5-4.5) | 2.73± 0.89 | 2.59 (1-4.77) | t=-0.101 p=0.919 |
| MSS AT. | 2.41± 0.63 | 2.27 (1.36-3.91) | 2.79± 0.88 | 2.77 (1.05-4.68) | t=2.761p= <b>0.007</b> |
| Analysis* (in-group) | t=5.898 <b>p&lt;0.001</b> | | t=-0.728 p=0.470 | | |

<sup>\*</sup> Dependent Sample t-test, \*\* Independent Sample t test, p<0.05 Statistically Significant, BT: Before Training Eğitim AT: After Training

Table 5. The Distribution of the Findings of the Relationship Between the HLSBS II and the MSQ Total Scale Score Averages (n=128).

| | | Negative Impact. | | | |
|---|---|---|---|---|---|
| | | Somatic Complaints BT. | Pain Symptoms | Coping Methods | MSQ |
| Health Responsibility | r | 0.146 | 0.171 | 0.088 | 0.163 |
| | р | 0.100 | 0.054 | 0.324 | 0.066 |
| Physical Activity | | 0.006 | 0.038 | -0.017 | 0.014 |
| | р | 0.947 | 0.666 | 0.853 | 0.878 |
| Nutrition | | -0.025 | 0.036 | 0.079 | 0.011 |
| | р | 0.782 | 0.686 | 0.378 | 0.898 |
| Spiritual Development | | 0.015 | 0.073 | 0.131 | 0.058 |
| | р | 0.868 | 0.411 | 0.140 | 0.514 |

| Interpersonal Relations | r | .186* | 0.097 | 0.169 | .178* |
|-------------------------|---|-------|--------|-------|-------|
| | р | 0.035 | 0.277 | 0.057 | 0.044 |
| Stress Management | r | 0.043 | -0.015 | 0.101 | 0.040 |
| | р | 0.629 | 0.867 | 0.258 | 0.653 |
| HLSBS II | r | 0.088 | 0.094 | 0.123 | 0.108 |
| | р | 0.326 | 0.290 | 0.166 | 0.224 |

<sup>\*</sup>r:Pearson Correlation Coefficient,p<0.05 Statistically Significant.

## Table 1. Research Workflow

## PRELIMINARY PROCESS

Obtaining permissions for scales, Literature research, Preparation of training program, Receiving expert opinions, Obtaining the permissions of the ethics committee and institution,

## IMPLEMENTATION STAGE

## (9,10,11. Class Student)

Sample creation: Taking the height and weight, body mass indexes of 1300 female students and reaching the sample group. Obtaining family and individual consent

